CLINICAL TRIAL: NCT03048448
Title: An Open-label, Single-dose, Parallel-group Study to Assess the Pharmacokinetics of Fevipiprant (QAW039) in Patients With Hepatic Impairment Compared to Matched Healthy Subjects
Brief Title: Pharmacokinetics of Fevipiprant (QAW039) in Patients With Hepatic Impairment Compared to Matched Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CQAW039A2108
Record Dates: First submitted 2017-01-27; First posted 2017-02-09 (Estimated); Last update posted 2020-12-11 (Actual); Status verified 2020-04

CONDITIONS: Hepatic Impairment
Keywords: Hepatic impairment,; Fevipiprant,; adults,; pharmacokinetics
MeSH Terms: interventions — fevipiprant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Fevipiprant 450mg (Experimental): 450mg Film Coated Tablet
  Interventions: Drug: Fevipiprant

INTERVENTIONS:
Drug: Fevipiprant — Single 450mg dose
  Other Names: QAW039

SUMMARY:
This study will characterize the pharmacokinetics (PK) of QAW039 after a single oral dose of QAW039 in patients with hepatic impairment compared to healthy matched control subjects.

DETAILED DESCRIPTION:
The purpose of this study is to determine if the pharmacokinetic profile of Fevipiprant is different in patients with hepatic impairment compared to healthy matched volunteers to an extent that would require an adjustment of the dosage. Data from this study will be used to guide enrollment criteria in future clinical trials and to support regulatory submission and labeling information.

ELIGIBILITY:
Inclusion Criteria:

All subjects

- Weight of at least 50 kg and no more than 120 kg and have a body mass index in the range 18.0-36.0 kg/m2

Patients with hepatic impairment

* Moderate hepatic impairment (Group 1): Child-Pugh Class B (7-9 points),
* Severe hepatic impairment (Group 2): Child-Pugh Class C (10-15 points
* Mild hepatic impairment (Group 4): Child-Pugh Class A (5-6 points)

Healthy subjects

* Match in age (±5 years), gender, smoking status, and weight (± 15%) to an individual patient.
* In good health as determined by past medical history, physical examination, electrocardiogram, laboratory tests and urinalysis at screening.

Exclusion Criteria:

All subjects

* History of hypersensitivity and/or idiosyncracies to QAW039 or to drugs of similar classes (CRTh2 antagonists).
* Use of co-medications that may impact QAW039 exposure such as broad range UGT inhibitors or strong inhibitors of OAT3, OATP1B3, and P-gp, including but not limited to probenecid, ritonavir, valproic acid, and rifampin
* Surgical or medical condition which might significantly alter the absorption, distribution, metabolism, or excretion of drugs, or which may jeopardize the subject in case of participation in the study.
* History of malignancy of any organ system (other than localized basal cell carcinoma of the skin), treated or untreated, within the past 5 years, regardless of whether there is evidence of local recurrence or metastases.
* Pregnant or nursing (lactating) women.
* Women of child-bearing potential

Patients with hepatic impairment

* Hepatic impairment due to non-liver disease (e.g., right heart failure)
* Current symptoms or history of encephalopathy Grade III or IV within the past 6 months
* Primary biliary liver cirrhosis and biliary obstruction
* Emergency room visit or hospitalization due to liver disease within the preceding 3 months.
* Severe complications of liver disease within the preceding 3 months.

Healthy subjects

* Liver disease or liver injury as indicated by abnormal liver function tests.
* Any single parameter of ALT, AST, γ-GT, alkaline phosphatase or serum bilirubin must not exceed 1.5 x upper limit of normal (ULN)
* Any elevation above ULN of more than one parameter of ALT, AST, γ GT, alkaline phosphatase or serum bilirubin will exclude a subject from participation in the study
* A positive Hepatitis B surface antigen or Hepatitis C test result.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2017-05-31 (Actual); Primary Completion 2019-04-22 (Actual); Study Completion 2019-04-22 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics: Plasma concentration of Fevipiprant by AUClast | 120 hours post-dose
  AUClast is the area under the plasma concentration-time curve from time zero to the time of the last quantifiable concentration
Pharmacokinetics: Plasma concentration of Fevipiprant by AUCinf | 120 hours post-dose
  AUCinf is the area under the plasma concentration-time curve from time zero to infinity
Pharmacokinetics: Plasma concentration of Fevipiprant by Cmax | 120 hours post-dose
  Cmax is the observed maximum plasma concentration following drug administration

SECONDARY OUTCOMES:
Relationship between plasma pharmacokinetics of Fevipiprant by AUClast and baseline hepatic function. | 120 hours post-dose
  AUClast (the area under the plasma concentration-time curve from time zero to the time of the last quantifiable concentration ) related to Child Pugh score
Relationship between plasma pharmacokinetics of Fevipiprant by AUCinf and baseline hepatic function. | 120 hours post-dose
  AUCinf (the area under the plasma concentration-time curve from time zero to infinity) related to Child Pugh score
Relationship between plasma pharmacokinetics of Fevipiprant by Cmax and baseline hepatic function. | 120 hours post-dose
  Cmax is the observed maximum plasma concentration following drug administration related to Child Pugh score
Pharmacokinetics of the metabolite CCN362 by AUClast | 120 hours post-dose
  AUClast is the area under the plasma concentration-time curve from time zero to the time of the last quantifiable concentration
Pharmacokinetics of the metabolite CCN362 by AUCinf | 120 hours post-dose
  AUCinf is the area under the plasma concentration-time curve from time zero to infinity
Pharmacokinetics of the metabolite CCN362 by Cmax | 120 hours post-dose
  Cmax is the observed maximum plasma concentration following drug administration

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (2):
- United States (2):
  - Novartis Investigative Site, Anaheim, California
  - Novartis Investigative Site, Orlando, Florida

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Results for CQAW039A2108 from the Novartis Clinical Trials Website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=17633
- See also: A Plain Language Trial Summary is available on novartisclinicatrials.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=516